CLINICAL TRIAL: NCT05507931
Title: A Pilot Feasibility Study to Develop a Broccoli Sprouts-enriched Diet in the Management of Ulcerative Colitis
Brief Title: Broccoli Sprouts for Mild Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Maine (Other)
Responsible Party: Principal Investigator, Grace Chen, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00210637; 2022-67017-36303 (Other Grant/Funding Number: USDA National Institute of Food and Agriculture (NIFA))
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Chronic Mild
Keywords: sulforaphane; inflammatory markers; Inflammatory bowel disease; diet; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 Serving of broccoli sprouts (Experimental): 113 grams
  Interventions: Dietary Supplement: 1 Serving of broccoli sprouts
- 3 Servings of broccoli sprouts (Experimental): 339 grams
  Interventions: Dietary Supplement: 3 Servings of broccoli sprouts

INTERVENTIONS:
Dietary Supplement: 1 Serving of broccoli sprouts — Participants will take 1 serving of broccoli sprouts daily for 28 days. The sprouts will be provided by the study team along with instructions on how to prepare the steamed broccoli sprouts (i.e., steamed for 10 minutes). In addition to taking the sprouts, participants will be asked to complete food diaries and surveys, collect blood and stool samples, as well as having 2 in-person visits.
  Arms: 1 Serving of broccoli sprouts
Dietary Supplement: 3 Servings of broccoli sprouts — Participants will take 3 servings of broccoli a day for 28 days. The sprouts will be provided by the study team along with instructions on how to prepare the steamed broccoli sprouts (i.e., steamed for 10 minutes). In addition to taking the sprouts, participants will be asked to complete food diaries and surveys, collect blood and stool samples, as well as having 2 in-person visits.
  Arms: 3 Servings of broccoli sprouts

SUMMARY:
The goal of this study is to determine the number of servings of broccoli sprouts sufficient to (1) increase sulforaphane levels in the stool and blood and (2) reduce inflammatory markers in patients with mild ulcerative colitis. This is a pilot feasibility study to prepare for a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Documented endoscopic diagnosis of ulcerative colitis
* Currently being treated with a stable dose of 5-ASAs, steroids, or any other medication approved for ulcerative colitis

  * If on 5-ASA, no dose changes within 2 weeks before the Day 0 visit
  * If on steroids, prednisone dose not more than 20 mg daily and entocort not more than 9 mg daily, with no dose changes within 2 weeks before the Day 0 visit
  * All other medications require a stable dose for at least 8 weeks prior to enrollment.
  * No dose changes to any IBD medication anticipated for the duration of the study
* Body Mass Index (BMI) values 18.5-40 kg/m2
* Not on total parenteral nutrition (TPN) or receiving tube feeds.
* Ability to understand the study procedures, benefits and risks, and sign a written informed consent document.
* Able to fill out questionnaires regarding dietary intakes, bowel symptoms, and study experience

Exclusion Criteria:

* Taking Non-steroidal anti-inflammatory drugs (NSAIDs)
* Following a medically-prescribed diet, on Total parenteral nutrition (TPN), or tube feeds
* Newly diagnosed (within past month), or uncontrolled diabetes or cardiovascular disease
* Antibiotics in the previous 2 weeks
* Consumption of more than 5 ½ cups of servings/day of fruits and vegetables as assessed by the National Cancer Institute (NCI) Diet History Questionaire III online Food Questionnaire.
* A known allergy or sensitivity to cruciferous vegetables like arugula, bok choy, broccoli, cabbage, cauliflower, or collard greens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of adopting a steamed broccoli diet in patients with ulcerative colitis as measured by self report of difficulty eating broccoli sprouts. | Day 28
  Self report documented in the end of study questionnaire. The questionnaire has 11 questions with the feasibility specifically linked to question 7, "how difficult was it to eat broccoli sprouts?" The answers range from 'not at all' (1) to 'very hard' (5) on a likert like scale.
Feasibility of adopting a steamed broccoli diet in patients with inflammatory bowel disease ulcerative colitis as measured by participant compliance. | Day 28
  Compliance is collected through self-report of the number of servings consumed.
Levels of sulforaphane in the stool | Day 28
  Level recorded in micrograms/gram.
Levels of sulforaphane in the blood | Day 28
  Level recorded in micrograms/gram.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Chen, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT05507931/ICF_000.pdf